CLINICAL TRIAL: NCT05016973
Title: A Clinical Study of RC48-ADC Combined With Triplizumab as Neoadjuvant Therapy Before Radical Resection of Myometrial Invasive Bladder Cancer
Brief Title: A Clinical Study of RC48-ADC Combined With Triplizumab For Treatment of Myometrial Invasive Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUNU-UC-102
Record Dates: First submitted 2021-07-25; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — disitamab vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC+ Triplizumab (Experimental): RC48-ADC on days 1 every 21 days plus triplizumab on days 1 every 21 days
  Interventions: Drug: RC48-ADC; Drug: Triplizumab

INTERVENTIONS:
Drug: RC48-ADC — 2.0mg/kg, Intravenous drip on days 1 every 21 days
  Other Names: Disitamab vedotin
Drug: Triplizumab — 240mg, Intravenous drip on days 1 every 21 days

SUMMARY:
The purpose of this project is to explore whether Monoclonal Antibody-MMAE Conjugate for Injection (RC48-ADC) combined with Triplizumab as a preoperative neoadjuvant therapy for myometrial invasive bladder cancer (MIBC) can achieve a good tumor descending period, so as to prolong disease-free survival and overall survival.

DETAILED DESCRIPTION:
Bladder cancer is the most common malignant tumor of the urinary system, mainly urothelial cancer, and its morbidity and mortality are increasing year by year. According to cancer statistics published by CACancerJClin, there were about 81000 new cases of bladder cancer in China in 2015, and the number of deaths from bladder cancer reached 33000. According to the depth of invasion, bladder cancer can be divided into superficial bladder cancer and muscular invasive bladder cancer. More than 70% of superficial bladder cancers recur after initial treatment, and about 15% eventually develop into invasive cancer. The prognosis of superficial bladder cancer is good (the 5-year survival rate is more than 90%). After entering the stage of myometrial invasion, the 5-year survival rate is only 60%, while the 5-year survival rate of patients with local advanced stage or metastasis is less than 15%.

Bladder cancer has been shown to be sensitive to chemotherapeutic drugs such as platinum, gemcitabine, doxorubicin and taxanes. The results show that in the stage of localized myometrial invasive bladder cancer, cisplatin-based neoadjuvant chemotherapy can significantly improve the median survival time of patients with myometrial invasive bladder cancer up to 31 months, showing a significant survival advantage.

Therefore, neoadjuvant chemotherapy is routinely recommended before radical resection for bladder cancer patients who can tolerate cisplatin. However, a single neoadjuvant chemotherapy can not meet the needs of all bladder cancer patients, so it is necessary to find new treatments to further supplement or improve the traditional neoadjuvant chemotherapy, so as to improve the postoperative survival of patients.

Since 2020, our group has also carried out a phase II clinical study of Tripril combined with GC regimen as a neoadjuvant regimen before MIBC. Triplet monoclonal antibody injection (Tuoyi) is a new type of recombinant humanized anti-PD-1 monoclonal antibody independently developed in China. At present, 18 cases have been enrolled in the study, 13 cases have been completed, and the rate of PaR and 31% pCR has reached 69.2%. The effect is similar to that of similar studies abroad. In spite of this, the combined therapy of immunity and chemotherapy is limited by the strong toxicity of platinum drugs, and some patients are still unable to tolerate it.

In recent years, the emergence of antibody drug conjugates (antibody-drugconjugate,ADC) provides a new choice for these patients. Studies have shown that ADC drugs and ICI drugs are highly complementary and safe. In addition, according to the results of the EV103 study, it can be found that the combination of ADC and ICI has a significant synergistic effect and has a strong and rapid shrinking effect on urothelial cancer. At the same time, these two drugs do not require high renal function, so they are very suitable for neoadjuvant therapy before MIBC.

RC48-ADC (Recombinant humanized Anti-HER2 Monoclonal Antibody-MMAE Coupling Agent for injection, referred to as RC48-ADC) independently developed by Rongchang Biopharmaceuticals in China is the first clinically approved HER2 antibody coupling drug in China. RC48-ADC exerts its anti-tumor effect through two main pathways: one is to interfere with cell transcription, growth and proliferation by inhibiting downstream signal pathways activated by HER2 (such as PI3K/AKT), and the other is the interference of microtubule formation by small molecule MMAE, which is mainly manifested by depolymerizing microtubules and inducing cell cycle arrest in G2max M phase. In addition, in vitro studies have shown that RC48-ADC has a tumor inhibitory effect on HER2 overexpressed cancer cells through antibody-dependent cell-mediated cytotoxicity (ADCC). About 25-30% of bladder cancers show high expression of HER2, and these tumors tend to have higher stage and grade, are more prone to invasion and metastasis and have a poor prognosis. Therefore, RC48-ADC has a high application prospect in bladder cancer with high expression of HER2.

The RC48-C005 study is a single-arm, open, multicenter II phase clinical study in China to evaluate RC48-ADC in the treatment of locally advanced or metastatic bladder urothelial carcinoma with overexpression of HER2. Through this study, it can be found that RC48-ADC has significant therapeutic efficacy and good safety in advanced urothelial cancer with high expression of Her-2.

Based on this, this study intend to use the combination of ADC drugs and ICI drugs (RC48-ADC combined with triplizumab) as preoperative neoadjuvant therapy for patients with high expression of MIBC in HER2, in order to achieve a better effect of tumor decline, so as to prolong the disease-free survival and overall survival of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with myometrial invasive bladder cancer are prepared for radical cystectomy;
2. HER2 overexpression confirmed by pathological biopsy: IHC2+ or IHC3+; subjects can provide tumor samples detected by HER2;
3. Age ≥ 18 years old and ≤ 80 years old;
4. Tumor clinical stage is (c) T2-3bN0M0;
5. ECOG score ≤ 1;
6. Subjects have not received systemic chemotherapy, ADC drugs or immunotherapy.
7. The important laboratory examination indexes meet the following requirements:

   1. Hemoglobin ≥ 90g/L.
   2. Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L.
   3. Platelet ≥ 100 × 109 / L.
   4. 3.5mmol/L ≤ serum potassium ≤ 5.5mmol/L.
   5. Liver function index: ALT, AST ≤ 1.5 times the upper limit of normal value (ULN), TBIL ≤ 1.5ULN.
   6. eGFR ≥ 50 mL/min
   7. The left ventricular ejection fraction (LVEF) was 50%.
   8. Subjects with serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CrCl) ≥ 50mL/min
8. The subject is volunteer to participate, and the subject must signed an informed consent form (ICF), indicating that it understands the purpose of this study and the required procedures, and is willing to participate in the study. Subjects must be willing and abide by prohibition and restrictions specified in the research program
9. Female subjects should be surgically sterilized or postmenopausal, or agree to use at least one medically approved contraceptive method (such as intrauterine device, contraceptive or condom) during the study treatment and within 6 months after the end of the study treatment period. The blood pregnancy test must be negative within 7 days before the study, and it must be non-lactation. Male subjects should agree to use at least one medically approved contraceptive method (such as condoms, abstinence, etc.) during the study treatment period and within 6 months after the end of the study treatment period.
10. Subjects are willing and able to follow the trial and follow-up procedures

Exclusion Criteria:

1. Patients who cannot tolerate radical cystectomy;
2. patients with myometrial invasive urothelial carcinoma with distant metastasis (abdominal CT scan + enhancement, chest CT scan, ECT- bone scan, PET-CT, MRI, etc.).
3. Uncontrollable concomitant diseases, including, but not limited to, persistent infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, arrhythmia, interstitial lung disease, severe chronic gastrointestinal disease associated with diarrhoea, or mental illness / social conditions, which will limit compliance with research requirements, significantly increase the risk of AE or impair the patient's ability to write informed consent.
4. Patients with drug allergy or hypersensitivity, patients with autoimmune diseases;
5. Received antineoplastic therapy within 3 weeks before the start of the study, including chemotherapy, radiotherapy, targeted therapy, immunotherapy and clinical research antineoplastic drug therapy.
6. Had received live attenuated vaccine or had serious infection or planned to receive any vaccine during the study period one month before entering the group.
7. Systemic corticosteroids or other systemic immunosuppressive drugs are used within 2 weeks before enrollment, or systemic immunosuppressive drugs are expected to be needed during the trial;
8. Serovirological examination (based on the normal value of the research center):

   HBsAg or HBcAb test results are positive, while HBVDNA copies are positive; HCVAb test results are positive (only if the PCR test result of HCVRNA is negative).

   The results of HIVAb test were positive.
9. Heart failure classified as grade 3 or above by the New York College of Cardiology (NYHA);
10. Active or progressive infections that require systematic treatment, such as active pulmonary tuberculosis;
11. Systemic diseases that have not been stably controlled by researchers, including diabetes, hypertension, liver cirrhosis, interstitial pneumonia, obstructive pulmonary disease, etc.
12. Serious arteriovenous thrombosis or cardio-cerebrovascular accidents occurred within 1 year before administration, such as deep venous thrombosis, pulmonary embolism, cerebral infarction, cerebral hemorrhage, myocardial infarction, etc., except for lacunar infarction that is asymptomatic and does not require clinical intervention;
13. Previous allogeneic hematopoietic stem cell transplantation;
14. Previous antibody-coupled drug therapy;
15. Pregnant or lactating women.
16. Suffering from any other disease, abnormal metabolism, abnormal physical examination or abnormal laboratory examination, according to the researchers, there is reason to suspect that the patient has a disease or condition that is not suitable for the use of research drugs, or will affect the interpretation of the results of the study, or put the patient at high risk;
17. Other situations that some researchers believe are not appropriate to participate in this study.

Elimination standard

1. Received other local or systemic treatments at the same time;
2. The simultaneous use of other foods and drugs that affected the judgment of tolerance; (3) In violation of the requirements of the study scheme, drugs were not given according to the dose and course of treatment specified in the study scheme;

(4) The quality of data recording was poor and the data was incomplete and inaccurate.

Termination criteria

1. Subjects asked to stop using the research therapy.
2. Recurrence (local, regional or distant).
3. For any clinical AE, laboratory examination abnormalities or concomitant diseases, according to the judgment of the researchers, continuing to participate in the study is not the greatest benefit to the subjects.
4. The researcher terminated the study.
5. The informed consent form can no longer be freely signed because of crime or forcible detention for the treatment of mental illness or physical illness (such as infectious diseases).
6. The adverse events and severity of other clinical trials of this study or study drugs suggest that the risk of the subjects is too high to continue the study;
7. The speed of enrollment in the research center is too slow to complete the enrollment plan within a limited time;
8. The quality of the clinical data is not good enough to continue the follow-up study;
9. The study is terminated due to the regulatory requirements or policy changes of the national drug administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Pathological response (PaR) rate per central pathology review | Up to approximately 6 months

SECONDARY OUTCOMES:
The pathological complete response rate refers to all target lesions disappear. | Up to approximately 6 months
  PCR (Pathological complete response rate) refers to all target nidus disappeared and repeated measurement evaluation at 4 weeks after RC.
Progression free survival: Follow-up was made after the first month after the operation, and then with an every three months until the tumor relapsed or progress. | Up to approximately 48 months
  PFS (Progression free survival) means from the random date to the first time disease progress or any cause of death, with the first appearance.
OS (Overall survival): The time from start of study treatment to date of death due to any cause. | Up to approximately 48 months
  OS (total survival time) refers to the total survival time of the subjects who survived at the last follow-up from the random date to the date of death of any cause. The total survival time of the subjects who were still alive at the last follow-up was deleted as the data of the last follow-up time. The overall survival time of the subjects who lost follow-up was recorded as data deletion according to the last confirmed survival time before the loss of follow-up. The total lifetime of data deletion is defined as the time from random grouping to deletion.
Adverse reaction rate: from the beginning of the study subjects receiving treatment, the adverse reactions caused by the treatment were recorded in detail. The adverse events that have not disappeared after chemotherapy should be followed up. | Up to approximately 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided